CLINICAL TRIAL: NCT01198860
Title: Tenofovir Disoproxil Fumarat - Phyllanthus Urinaria- Adenosma Glutinosum - Eclipta Prostrata - Ascorbic Acid is Effective in the Long-term Treatment of Chronic and Acute Hepatitis B.
Brief Title: Treatment on HBeAg Positive or HBeAg Negative in Chronic Hepatitis B
Acronym: HBV
Status: Approved for marketing | Type: Expanded Access
Sponsor: Nguyen Thi Trieu, MD (Individual)
Responsible Party: Sponsor-Investigator, Nguyen Thi Trieu, MD, Trần Minh Đức, Trieu, Nguyen Thi, M.D.
Organization: Trieu, Nguyen Thi, M.D. (Individual)
Other Study IDs: HBsAg 07-10 - Private Clinic
Record Dates: First submitted 2010-09-04; First posted 2010-09-10 (Estimated); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: CHRONIC HEPATITIS B
Keywords: HBsAg
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Ascorbic Acid; Tenofovir

INTERVENTIONS:
Drug: CTH Chronic Hepatitis B — Drug:
  * Tenofovir
  * Phyllanthus Urinaria
  * Adenosma Glutinosum
  * Eclipta Prostrata
  * Ascorbic Acid
  Other Names: - Ascorbic Acid; - Phyllanthus Urinaria; - Adenosma Glutinosum; - Eclipta Prostrata; - Tenofovir

SUMMARY:
Phyllanthus Urinaria - Adenosma Glutinosum - Eclipta Prostrata - Ascorbic Acid combination plus Tenofovir in treatment of acute and chronic hepatitis B. Method the combination of drugs derived from natural and artificial medicaments.

Has stronger effect on immune system, effective good against HBV replication. This is a substantial new insight into the pathogenesis of disease, with a clear path toward clinical application, or which would lead to a substantial advance and perfect in management or public health policy.

DETAILED DESCRIPTION:
Recent studies have proved Phyllanthus Urinaria - Adenosmatis Glutinosum - Eclipta Prostrata - Ascorbic Acid combination plus Tenofovir in treatment of acute and chronic hepatitis B. Method the combination of drugs derived from natural and artificial medicaments. To made a clean jobs for HBV - DNA in the patient's body - hope this is a new step of medicine, will no longer exist phrase "chronic HBV infection " Methods of safety, therapeutic effect on expected cost savings should easily apply to everyone everywhere in the world. According to the investigation and must be called , Chronic HBV infection is an important worldwide cause of morbidity, mortality and source of potential new infections. There are an estimated 350 million carriers of HBV in the world. In China, Southeast Asia and sub-Saharan Africa, as many as 10-15% of the population are chronically infected. In North America and Northern Europe, infection and carrier rates are much lower, usually below 1%. Intermediate carrier rates of 1-5% are found in Southern Europe (e.g., Italy, Greece and Spain), parts of South and Central America, the Middle East and Japan. Persistent infection develops in over 90% of perinatally infected children and in 3-10% of people who become infected after the age of 6 years. Worldwide, it has been estimated that more than one million people die annually due to HBV-related end stage diseases such as cirrhosis and hepatocellular carcinoma.

The goal of antiviral therapy for hepatitis B is to reduce a patient's risks for progressive liver disease through prolonged suppression and eradication of HBV infection and to arrest or ameliorate HBV-related liver damage.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* Males and females ≥ 18 years of age with chronic and acute hepatitis B.
* Hepatitis B surface antigen (HBsAg)(+) for a minimum of 6 months prior to entry.
* Hepatitis B envelope antigen (HBeAg)(+) or (-) at baseline.
* Patients having treated or untreated
* Patients with compensated liver function (Child-Pugh score ≤ 6).
* Informed writted consent.

Exclusion Criteria:

* Any serious or active medical or psychiatric illness which, in the opinion of the investigator, would interfere with patient treatment, assessment or compliance with the protocol. or cytokine-based therapies with possible activity in hepatitis B disease within 6 months prior to study screening.
* Organ or bone marrow transplant recipients.
* Evidence of active liver disease to operate.
* Received immunoglobulins, interferon or other immune e to other causes (e.g., Wilson's disease, hemochromatosis, autoimmune hepatitis, hepatitis C, hepatitis D or HIV.)
* Patients taking parenteral (intravenous or intramuscular or subcutaneous) or oral steroids, immuno-suppressant therapies or chemotherapeutic agents within 2 months of study screening or expected to receive these agents during the course of the study.
* Clinically relevant alcohol or drug use or history of alcohol or drug use considered by the investigator to be sufficient to hinder compliance with treatment, follow up procedures or evaluation of adverse events.
* Hepatocellular carcinoma.
* Serious concurrent medical illness other than hepatitis B.
* History of hypersensitivity to nucleoside analogues.
* Women of childbearing potential not practising adequate contraception.
* Pregnancy or lactation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Nguyễn Thị Triệu, Dr., Study Director — Tran Minh Duc, Dr.
Locations (2):
- Saigon Biopharma LLC, Wilmington, Delaware, United States
- Saigon Biopharma Company Limited, Hồ Chí Minh, Ho Chi Minh City, Vietnam